CLINICAL TRIAL: NCT02926209
Title: Post Market Evaluation of Aer-O-Scope Visualization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Further development needed to facilitate easier polypectomy - device improvement
Sponsor: GI View Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 934CLD
Record Dates: First submitted 2016-09-27; First posted 2016-10-06 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: colonoscopy; adenoma; polyp; crc screening
MeSH Terms: conditions — Neoplasms; Adenoma; Polyps | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aer-O-Scope First (Active Comparator): Patients in this arm will undergo colonoscopy using the Aer-O-Scope followed by colonoscopy using a conventional colonoscope
  Interventions: Device: Aer-O-Scope (Colonoscopy); Procedure: Colonoscopy (Conventional Colonoscope)
- Conventional Colonoscope First (Active Comparator): Patients in this arm will undergo colonoscopy using a conventional colonoscope followed by colonoscopy using the Aer-O-Scope
  Interventions: Device: Aer-O-Scope (Colonoscopy); Procedure: Colonoscopy (Conventional Colonoscope)

INTERVENTIONS:
Device: Aer-O-Scope (Colonoscopy) — Patients in the "Aer-O-Scope first arm" will undergo a colonoscopy with the Aer-O-Scope, removing any polyps detected, followed by a colonoscopy using a conventional colonoscope, removing any polyps not previously detected with the Aer-O-Scope.
  Other Names: CRC Screening
Procedure: Colonoscopy (Conventional Colonoscope) — Patients in the "conventional colonoscope first arm" will undergo a colonoscopy with a conventional colonoscope, removing any polyps detected, followed by a colonoscopy using the Aer-O-Scope, removing any polyps not previously detected with the conventional colonoscope
  Other Names: CRC Screening

SUMMARY:
This will be a prospective multi-center, multi-national comparative non-blinded clinical investigation. Each subject will undergo back-to-back tandem colonoscopies with the Aer-O-Scope Colonoscope System and a conventional colonoscope since this is a tandem colonoscopy study, each subject will serve as their own control. The 1st procedure will be randomized, half to Aer-O-Scope Colonoscope System and half to conventional colonoscope. The same investigator will perform both procedures on each subject. All pathologies found will be either removed or tattooed. Unmarked pathologies found on second pass will represent those missed during the 1st pass, thus making the subject and the control one and the same. Tattooed pathologies that can be removed endoscopically will be removed in an additional colonoscopy. This may occur if a large polyp cannot be removed for any reason with the Aer-O-Scope, but can be removed with conventional colonoscopy.

DETAILED DESCRIPTION:
Subjects will be randomized in blocks of twenty (20) for either Aer-O-Scope or conventional colonoscopy as the first procedure. Physicians will be notified of the procedural order immediately prior to first colonoscopy. Up to the first ten (10) cases for each physician (system operation training cases) will all begin with the Aer-O-Scope colonoscopy as the first procedure.

The primary endpoint of AMR was chosen as this measure appears to be related to the performance of colonoscopy and reduction in colorectal cancer incidence. During the course of the last decade, several major visualizations studies have been performed and it has become common practice to use the "second-pass" method for measuring colonoscopy visualization methods, iii, iv. In the "second-pass" method, during the course of the first colonoscopy, all visualized lesions are removed (or tattooed in the event that they cannot be removed for any reason.). Any unmarked abnormalities discovered during the second pass colonoscopy are considered to be missed pathologies for the first pass colonoscopy.

All endpoints related to timing will be measured using a stopwatch and overall time stamp from the Aer-O-Scope or conventional colonoscope. Time to perform therapeutic interventions with Aer-O-Scope as well as a description of said interventions will also be recorded. The same instruments will be used to measure all procedures and will be calibrated as dictated by the manufacturer.

All equipment used during the course of this clinical investigation will undergo calibration and testing as per the manufacturing instructions. The Aer-O-Scope Colonoscope System has an automated calibration system and diagnostic test that run daily. Conventional colonoscopes will be maintained as per hospital/manufacturer protocol.

Recruited subjects who are withdrawn as a result of poor bowel prep or any other medical determination leading to the inability to undergo colonoscopy and/or tandem colonoscopy will be replaced. A poor prep is defined as having a score of score of 0 or 1 in the Boston Bowel Preparation Scale (BBPS). The BBPS scores are as follows:

0 = Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.

1. = Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid.
2. = Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well.
3. = Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.

Any subject withdrawn as a result of physician discretion due to concomitant medical issues will be withdrawn prior to the actual colonoscopic procedures. Patients with a large polyp (>20mm) removed during the first pass with a conventional colonoscope will be withdrawn. Patients who receive treatment during the first pass with clips (no other option available) will be withdrawn.

Coagulation therapy should be performed either with Argon Plasma Coagulation (APC) or another cautery tool or contact thermal device as per clinical protocol. For the purpose of this clinical investigation, clips should not be used unless there is no alternative. Patients treated with clips prior to their final pass colonoscopy, will be withdrawn from the investigation.

Physicians may also withdraw any patient due to medical causes if deemed appropriate, including patients that have undergone at least one (1) procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is indicated for screening, diagnostic (minor complaints such as rectal bleeding or minor abdominal pain) or surveillance colonoscopy
2. Subject willing to undergo tandem colonoscopies with Aer-O-Scope Colonoscope and a conventional colonoscope (including a single colon preparation bowel cleansing)
3. Subject between the ages of 45 and 75 (patients between the ages of 45 and 50 must have a family history of a first degree relative with onset of colon cancer before the age of 60).
4. Subject is able to understand and willing to sign informed consent form

Exclusion Criteria:

1. Personal history of colorectal neoplasia including familial adenomatous polyposis or hereditary nonpolyposis, colon cancer (HNPCC).
2. Diagnosis of active (flaring) inflammatory bowel disease (active ulcerative colitis or Crohn's colitis), bowel obstruction, or acute diverticulitis, or known severe diverticulosis, fecal incontinence or any known large-bowel disease that would require a predetermined therapeutic colonoscopy (non-screening, non-diagnostic or non-surveillance cases)
3. Severe gastrointestinal tract-related symptoms, or complaints, suggesting performance of a pre-determined therapeutic colonoscopy (non-screening, non-diagnostic or non-surveillance cases)
4. History of colonic resection
5. Clinically significant cardiovascular or pulmonary disease.
6. Cancer or other life threatening disease or significant chronic condition that puts the subject at risk.
7. Blood-clotting disorders and/or current anticoagulant therapy (Subjects taking up to 100mg aspirin for prophylactic treatment are acceptable for this study)
8. Pregnancy
9. Previous radiation therapy to the abdomen
10. Morbid Obesity (BMI > 40 kg/m2)
11. Drug abuse or alcoholism
12. Subject is bed-ridden and/or unable to adequately communicate
13. Subject is under custodial care
14. Subject has a history of psychiatric disorders which would prevent compliance with study instructions
15. Participation in a clinical study within the previous 30 days

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Santo, MD, Principal Investigator — Tel Aviv Souraski Medical Center, Israel; Klaus Mergener, MD, PhD, MBA, Principal Investigator — Waldron Endoscopy Center, Tacoma, WA, USA
Locations (2):
- Waldron Endoscopy Center, Tacoma, Washington, United States
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 104 subjects were screened out of which 100 recruited into the study. Three (3) subjects were removed from the study by the physician during the procedures for medical reasons and one (1) subject did not complete the bowel preparation and was therefore excluded. One (1) subject withdrew consent prior to the procedure.
Period: Study Cohort
Arm/Group | Aer-O-Scope First | Conventional Colonoscope First
Started | 42 (Training cohort patients Aer-O-Scope as first followed by a conventional colonoscopy) | 37
Completed | 41 | 37
Not Completed | 1 | 0
Not completed — Poor Bowel Preparation | 1 | 0
Period: Training Cohort - First Patients
Arm/Group | Aer-O-Scope First | Conventional Colonoscope First
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: These patients were part of the physician training cohort. The first 10 subjects for each physician constitute this cohort
Groups:
- Training Cohort: The first 20 subjects in this study were in the training cohort which was not evaluated statistically for the objectives.
Arm/Group | Training Cohort
Number analyzed (Participants) | 98
Age, Customized [Mean (Standard Deviation); unit: years] — Population of participants Population: The first 20 participants were in the training cohort and were therefore not analyzed.
  years
    Overall Total Subjects | 55.41 (5.84)
    Study Cohort: number analyzed (Participants) | 78
    Study Cohort | 55.33 (5.99)
Sex: Female, Male [Count of Participants; unit: Participants] — 58 male and 40 female
  Participants
    Female | 40
    Male | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 98

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Miss Rates
Description: Determined by second pass colonoscopy - lesions detected in second pass represent lesions missed during first pass - adenomatic status based on histopathology.
  Three (3) lesions were missed by the Aer-OScope and detected with the subsequent conventional colonoscopy. Two (2) polyps were not removed and an additional one (1) was not retrieved.
  Data was missing for two (2) lesions by the Conventional Colonoscopy (CC)
Time Frame: Through study completion, an average of one year
Measure: Number; unit: missed adenomas
Arm/Group | Aer-O-Scope First | Conventional Colonoscope First
Number analyzed (Participants) | 41 | 37
missed adenomas | 3 | 2

2. Secondary Outcome: Polyp Miss Rates (PMR) for Each Study Arm
Description: Determined by second pass colonoscopy - lesions detected in second pass represent lesions missed during first pass
Time Frame: Through study completion, an average of one year
Measure: Number; unit: missed polyps
Arm/Group | Aer-O-Scope First | Conventional Colonoscope First
Number analyzed (Participants) | 41 | 37
missed polyps | 4 | 2

3. Secondary Outcome: Advanced Adenoma Miss Rates (AAMR) for Each Study Arm
Description: Determined by second pass colonoscopy - lesions detected in second pass represent lesions missed during first pass - adenomatic status based on histopathology.
Time Frame: Through study completion, an average of one year
Measure: Number; unit: missed advanced adenomas
Arm/Group | Aer-O-Scope First | Conventional Colonoscope First
Number analyzed (Participants) | 41 | 37
missed advanced adenomas | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study and 24 hours post procedure per patient
Description: Anticipated adverse device effects include bloating, flatulence mild in nature, ano-rectal fissures and minor discomfort. These symptoms are all transient and do not pose a potential risk to the subjects' health. These were listed as expected events and were not recorded
Groups:
- Training Cohort: The first 10 patients for each physician were considered the physician training cohort. These patients were not analysed with the final study cohort which included the Aer-O-Scope First and Conventional Colonscope First Arms. No adverse events, immediate or delayed occurred during the course of this study, as such, the arms were combined for reporting
- Aer-O-Scope First: Patients in this arm will undergo colonoscopy using the Aer-O-Scope followed by colonoscopy using a conventional colonoscope
  Aer-O-Scope (Colonoscopy): Patients in the "Aer-O-Scope first arm" will undergo a colonoscopy with the Aer-O-Scope, removing any polyps detected, followed by a colonoscopy using a conventional colonoscope, removing any polyps not previously detected with the Aer-O-Scope.
  Colonoscopy (Conventional Colonoscope): Patients in the "conventional colonoscope first arm" will undergo a colonoscopy with a conventional colonoscope, removing any polyps detected, followed by a colonoscopy using the Aer-O-Scope, removing any polyps not previously detected with the conventional colonoscope No adverse events, immediate or delayed occurred during the course of this study, as such, the arms were combined for reporting
- Conventional Colonoscope First: Patients in this arm will undergo colonoscopy using a conventional colonoscope followed by colonoscopy using the Aer-O-Scope
  Aer-O-Scope (Colonoscopy): Patients in the "Aer-O-Scope first arm" will undergo a colonoscopy with the Aer-O-Scope, removing any polyps detected, followed by a colonoscopy using a conventional colonoscope, removing any polyps not previously detected with the Aer-O-Scope.
  Colonoscopy (Conventional Colonoscope): Patients in the "conventional colonoscope first arm" will undergo a colonoscopy with a conventional colonoscope, removing any polyps detected, followed by a colonoscopy using the Aer-O-Scope, removing any polyps not previously detected with the conventional colonoscope No adverse events, immediate or delayed occurred during the course of this study, as such, the arms were combined for reporting
Arm/Group | Training Cohort | Aer-O-Scope First | Conventional Colonoscope First
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 0/20 | 0/40 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02926209/Prot_SAP_000.pdf